CLINICAL TRIAL: NCT02322528
Title: Evaluation of Ocular Surface Inflammatory Mediators and Ocular Surface Metrology Effected by Lotemax
Brief Title: Evaluation of Ocular Surface Inflammatory Mediators Effected by Lotemax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, James V. Aquavella, MD, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 47817
Record Dates: First submitted 2014-04-16; First posted 2014-12-23 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Sjogren's Disease
Keywords: Non-invasive instruments; Environment; Wavefront; Placido Disk; Ellipsometer; Thermal Imaging
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Administration of Lotemax (Other): An FDA approved drug (Lotemax) will be administered to both eyes to induce an inflammatory mediated response.
  Interventions: Drug: Administration of Lotemax

INTERVENTIONS:
Drug: Administration of Lotemax — An FDA approved drug (Lotemax) will be administered to induce an inflammatory mediated response in both eyes.

SUMMARY:
The purpose of this study is to evaluate the effects of an anti-inflammatory drug (Lotemax®) on the surface of the eye and tear film (a film that coats the eye which is made up of oil and water).

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 50-70
* Diagnosed with Sjogren's Disease
* Good general health (defined by medication use that has not changed within the last 2 months and the absence of medical conditions that are deemed confounding to the data as determined by the PI)
* Ability to give informed consent
* Willing to spend time for the study; approximately one hour for a screening visit and between 60-90 minutes for each of the measurement visits
* Either gender
* Any racial or ethnic origin

EXCLUSION CRITERIA:

* Use of any prescription ocular medication (such as but not limited to, glaucoma medications and Restasis) used within 14 days of the screening visit or started prior to the measurement visit(s).
* Current acute eye disease that affects the surface of the eye such as, but not limited to blepharitis, ocular allergy, and infection.
* Subjects who have had cataract surgery less than one year ago
* Use of soft or hard contact lenses.
* Female subjects may not be pregnant or lactating (subjects will be asked to self-report these conditions).
* Inability to provide analyzable data

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James V Aquavella, MD, Principal Investigator — University of Rochester
Locations (1):
- Flaum Eye Institute at the University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Administration of 0.5% Lotemax: An FDA approved drug (Lotemax) will be administered to both eyes to induce an inflammatory mediated response.
Period: Overall Study
Arm/Group | Administration of 0.5% Lotemax
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Administration of Lotemax
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (4.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Temperature of Both Eyes
Description: Lotemax® is an FDA-approved ophthalmic suspension for the treatment of steroid-responsive inflammatory conditions which include dry eye associated ocular surface inflammation. Lotemax® will serve as a vehicle to study the changes in the inflammatory mediators on the surface of the eye as well as collect the inflammatory mediators for laboratory analysis, utilizing Luminex instrumentation and standard ELISA assays.
Time Frame: baseline, 30 minutes, week 1, week 2
Measure: Mean (Standard Deviation); unit: degrees celcius
Arm/Group | Administration of 0.5% Lotemax
Number analyzed (Participants) | 10
degrees celcius
  baseline | 33.95 (0.13)
  30 minutes | 34.3 (0.13)
  week 1 | 33.93 (0.12)
  week 2 | 33.95 (0.13)

2. Primary Outcome: Visual Quality
Description: Using a Shack Hartmann wavefront sensor, measured root mean square of wavefront aberrations caused by dynamic tear film changes.
Time Frame: baseline, 30 minutes, week 1, week 2
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Administration of 0.5% Lotemax
Number analyzed (Participants) | 10
microns
  baseline | 0.48 (0.04)
  30 minutes | 0.54 (0.04)
  week 1 | 0.49 (0.08)
  week 2 | 0.48 (0.04)

ADVERSE EVENTS:
Arm/Group | Administration of 0.5% Lotemax
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes